CLINICAL TRIAL: NCT00222820
Title: Depression: The Search for Treatment-Relevant Phenotypes
Brief Title: Depression: The Search for Treatment-Relevant Phenotypes-Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Mental Health Intervention Research Center (MHIRC) (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 011015
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Interpersonal Psychotherapy

INTERVENTIONS:
Drug: escitalopram
Behavioral: Interpersonal Psychotherapy

SUMMARY:
We are doing this pilot study to learn more about four aspects of treating depression:

1. The features of a depressed person's mood and anxiety and how these features affect a person's capacity to get better and stay better.
2. If depressed people with certain features of mood and anxiety respond better to therapy, medication or a combination of therapy and medication.
3. Whether or not a person's personality traits affect how they respond to treatment.
4. The gene involved in processing antidepressant medication

DETAILED DESCRIPTION:
This pilot study is an experimental investigation designed so that consenting subjects are randomly assigned to pharmacotherapeutic or psychotherapeutic interventions for depression.

For the initial phase of treatment, subjects will be randomly assigned to treatment with an SSRI, (escitalopram oxalate or citalopram hydrobromide), or with interpersonal psychotherapy (IPT). Escitalopram will be prescribed for all patients randomized to the medication arm of the study, unless the study psychiatrist determines that citalopram is more clinically appropriate. Escitalopram and citalopram are FDA-Approved SSRI antidepressants indicated for the treatment of depression. In order to optimize outcomes and emulate usual clinical practice, subjects who do not meet response criteria (defined as a 50% reduction in baseline Hamilton Rating Scale for Depression [HRS-D]) or meet stabilization criteria (defined as a mean HRS-D < 7 for 3 weeks) at acute phase Visit 7 or Visit 13 of treatment will have the other treatment added. Subjects who meet stabilization criteria (mean HRS-D < 7 for 3 weeks) at any time between acute phase Visit 13 and 21 will enter the 6-month continuation phase and continue with the treatment that led to their stabilization. Subjects who have not met stabilization criteria by acute phase Visit 21 will remain in active treatment and be offered alternative pharmacotherapy. Subjects who have not responded by acute phase Visit 32 will be discontinued from the protocol and referred for alternative treatment and care.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 2 Age 18-65 3. Currently experiencing an episode of major depression 4. Not currently receiving effective treatment 5. Females of childbearing potential: practicing an acceptable form of birth control 6. Subjects with suicidal ideation are eligible as long as outpatient treatment is deemed safe 7. Willingness and ability to give informed consent.

Exclusion Criteria:

1. History of manic or hypomanic episodes;
2. History of schizophrenia or schizoaffective disorder;
3. Current primary diagnosis of anorexia nervosa or bulimia nervosa;
4. Current psychosis;
5. Drug and/or alcohol dependence or abuse within the past three months (episodic abuse related to mood episodes will not exclude a subject);
6. Antisocial personality disorder (other Axis II disorders will not be exclusionary);
7. Organic affective syndrome;
8. Renal or liver disease;
9. Epilepsy;
10. Cardiovascular disease;
11. Uncontrolled illnesses, including untreated hypertension or unstable endocrine diseases.
12. Women who are or are plan to become pregnant during the course of this study
13. Subjects who require inpatient treatment because of suicidal risk or psychosis
14. Subjects with a well-documented history of an inability to tolerate one of the study treatments or are currently receiving treatment with an effective antidepressant therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2002-04; Study Completion 2004-09

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression

SECONDARY OUTCOMES:
Inventory of Depressive Symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Frank, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychaitric Institute and Clinic, Pittsburgh, Pennsylvania, United States